CLINICAL TRIAL: NCT06963398
Title: A Phase 1 Study, Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of HS-10529 Monotherapy in KRAS G12D Patients With Advanced Solid Tumors
Brief Title: A Study of HS-10529 in KRAS G12D Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10529-101
Record Dates: First submitted 2025-04-29; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors; KRAS G12D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-10529 (Experimental)
  Interventions: Drug: HS-10529

INTERVENTIONS:
Drug: HS-10529 — Participants in all subjucts will receive HS-10529

SUMMARY:
HS-10529 is an oral, highly selective, small molecular inhibitor of KRAS G12D. This study will evaluate the safety, tolerability, pharmacokinetics and clinical activity of HS-10529 in KRAS G12D patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a phase 1, first-in-human, study of HS-10529, consisting of dose escalation and dose expansion, which is aimed to assess the safety and tolerability of HS-10529 in KRAS G12D patients with advanced solid tumors and evaluate the preliminary efficacy of HS-10529.

ELIGIBILITY:
Inclusion Criteria:

* At least age of 18 years at screening.
* Patients of advanced solid tumor，who have progressed on or intolerant to standard therapy.
* With measurable lesion according to RECIST 1.1.
* Agree to provide fresh or archival tumor tissue.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0~1.

Exclusion Criteria:

* Previous or current treatment with KRAS G12D inhibitors.
* Uncontrolled pleural, ascites or pericardial effusion.
* Known and untreated, or active central nervous system metastases.
* History of other primary malignant tumors.
* Serious, uncontrolled, or active comorbidities.
* Refractory nausea, vomiting, or chronic gastrointestinal diseases, or inability to swallow oral medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) or maximum applicable dose (MAD) | up to 24 months

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | up to 24 months
Plasma concentration of HS-10529 | up to 36 months